CLINICAL TRIAL: NCT04860128
Title: New Technologies as a Tool for Health Promotion in Schoolchildren of Compulsory Secondary Education: Effects of Sports Technology Applications on the Physical and Psychological Health of Adolescents
Brief Title: New Technologies as a Tool for Health Promotion in Schoolchildren of Compulsory Secondary Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Raquel Vaquero-Cristóbal, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CE022102
Record Dates: First submitted 2021-04-20; First posted 2021-04-26 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Adolescent Behavior; Physical Activity; New Technologies
Keywords: Adolescents; Physical activity; Psychology; New Technologies
MeSH Terms: conditions — Adolescent Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- "PACER" Application (Experimental): It is an application that allows the recording of the sports activities performed. It includes alerts and reminders that allow you to plan your sports practice in advance, as well as a weekly record of the activities and kilometers run, and a comparative analysis with the previous week.
  Interventions: Behavioral: Sports technology application
- "MapMyWalk" Application (Experimental): It is an application that promotes the practice of physical activity by recording the sports activities that the subject performs, as well as the dissemination of the same in social networks and participation in challenges available to users around the world. In addition, this application includes reminders of physical activity and personal achievements to encourage the practice of sports.
  Interventions: Behavioral: Sports technology application
- "Strava" Application (Experimental): It is an application that promotes sports practice, nutritional habits and the necessary rest. Nutrition and sleep will be introduced as variables that favor a healthy lifestyle.
  Interventions: Behavioral: Sports technology application
- "POKEMON GO" APPLICATION (Experimental): It is a mobile game that favors the increase of physical activity because it is necessary to walk to achieve the proposed objectives.
  Interventions: Behavioral: Sports technology application
- Control Group (No Intervention): They will not use any type of sports technology application. They will continue to perform their daily activities without intervention.

INTERVENTIONS:
Behavioral: Sports technology application — Each of the intervention groups will use in after-school hours a different mobile app for 12 weeks, with a frequency and duration of 60 minutes of training, at least three times a week. A weekly record will be kept by the adolescents in which they will have to indicate the weekly practice frequency, the duration of the activity and the kilometers covered through a report that the adolescents will deliver to the teacher at the end of each week.
  Arms: "MapMyWalk" Application; "PACER" Application; "POKEMON GO" APPLICATION; "Strava" Application

SUMMARY:
The rapid development of new technologies could be one of the causes that has favored changes in the lifestyle habits of young people. Research carried out to date shows that new technologies could be useful in increasing levels of physical activity and motivation to practice sports. However, these studies have major limitations that make it difficult to generalize the results.

The objectives of the present project are: 1) to determine the influence of the use of new technologies on the levels of sports practice and the physical and psychological health of adolescents; 2) to analyze the effects of a physical-sports activity program that integrates new technologies through mobile applications related to physical exercise on the level of physical activity and the physical and psychological health of adolescents; and 3) to analyze the adherence that this type of program generates in the medium term in adolescents as a function of age and gender.

The project will be divided into two phases. In the first phase, 500 students from the centers of Compulsory Secondary Education will be included, who will undergo physical tests, questionnaires related to sports practice and physical and psychological health, and an anthropometric assessment. In the second phase, an intervention will be carried out with four experimental groups and a control group. The four experimental groups will use different technological applications outside school hours for 12 weeks. Participants will keep a weekly record of physical activity and pre-, post and re-test measurements will be taken to evaluate the efficacy of the sports technology applications in increasing and maintaining physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Be a student of compulsory secondary education
* Not present any disease or surgical operation that would prevent the performance of the physical tests or the follow-up of the established intervention.
* Complete the questionnaires provided and carry out the established tests in their entirety
* Have access to any mobile device that allows access to the technological sports applications used in the intervention.

Exclusion Criteria:

* Failure to complete the questionnaires provided and/or to take the prescribed tests in their entirety
* Failure to complete scheduled intervention activities.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Use of internet (CERI Questionnaire) | Through study completion, an average of 1 year
  To measure the frequency of Internet use through new communication technologies, the CERI questionnaire (Fargues et al. 2009) will be used, which includes 10 questions rated on a scale of 1 to 4, with 1 being "almost never" and 4 "almost always".
Use of mobile phone (CERM Questionnaire) | Through study completion, an average of 1 year
  To measure the frequency of cell phone use, regardless of whether it is for social networks, video games, etc., the CERM questionnaire (Fargues et al. 2009) will be used, which includes 10 questions rated on a scale of 1 to 4, with 1 being "almost never" and 4 being "almost always".
Satisfaction with life (Life Satisfaction Scale) | Through study completion, an average of 1 year
  Life satisfaction is defined as a person's overall evaluation of his or her life. The person examines the tangible aspects of his or her life and compares them with a standard or criterion chosen by him or her, arriving at a judgment about satisfaction with his or her life (Pavot et al., 1991). Thus, judgments about satisfaction depend on the comparisons that the subject makes between the circumstances of his or her life and a standard that he or she considers appropriate. The life satisfaction scale (Diener et al., 1985) provides information on feelings of happiness, feelings of loneliness and satisfaction in school among adolescents, obtaining an overall assessment of life satisfaction. The scale is composed of five questions that are answered on a scale of 1 to 5, with 1 being "strongly disagree" and 5 "strongly agree". A higher score indicates greater satisfaction with life.
Physical Activity Level (International Physical Activity Questionnaire for Adolescents) | Through study completion, an average of 1 year
  The PAQ-A (Martínez-Gómez et al., 2009) will be used to establish the level of sports practice of the adolescents. This questionnaire includes eleven questions related to the practice of physical activity in school, after school, household chores and travel. The questionnaire makes it possible to classify adolescents as inactive or active (light, moderate or vigorous intensity).
Satisfaction of basic psychological needs (Psychological Need Satisfaction in Exercise Scale) | Through study completion, an average of 1 year
  Considering that the basic psychological needs are 3: competence, autonomy and social relationships, the Psychological Need Satisfaction in Exercise Scale (Wilson et al., 2006), composed of eighteen items (six for each of the dimensions) will be used to assess the degree of satisfaction with these basic psychological needs. For its completion, a scale of 1 to 6 will be used, with 1 being "totally false" and 6 "totally true".
Back pain (Nordic Questionnaire) | Through study completion, an average of 1 year
  Spinal pathologies, including back pain, are among the most common in recent decades, due to the lack of postural hygiene caused by postures maintained over time. Back pain refers to any of the areas that make up the back (cervical, dorsal, lumbar and shoulder areas). With the Nordic Questionnaire (Martínez and Alvarado, 2017), the aim is to obtain information on the regions in which adolescents present back pain. For this purpose, the questionnaire includes images that specify the place to which each region of the back refers, and questions related to the decrease in autonomy caused by pain in those regions.
Mediterranean Diet Quality (KIDMED Questionnaire) | Through study completion, an average of 1 year
  The KIDMED questionnaire (Serra-Majem et al., 2004) will be used to establish the level of adherence of adolescents to the Mediterranean diet. It consists of 16 questions that are scored with a value of -1 if they denote a negative connotation with respect to the Mediterranean diet, or with a +1 if they are positive in relation to the diet. The index ranges from 0 to 12 points and the results are classified as: optimal Mediterranean diet (>8 points), requires improvement to adjust intake to Mediterranean patterns (4-7 points), and very low diet quality (≤ 3 points). The questions included in the questionnaire are related to the main foods included in this type of diet (fruit, vegetables, bread, etc.).
Physical condition (Maximal oxygen consumption) | Through study completion, an average of 1 year
  The 20-m shuttle run test evaluates maximal aerobic capacity by means of an incremental 20-meter out-and-back test. The initial speed of the test is 8.5 km/h and is increased every minute by an audible signal. The test ends when the subject stops or fails to reach the reference line two consecutive times. The speed recorded is the speed reached in the last stage that the subject is able to complete. Through the equations of Leger, Mercier, Gadoury and Lambert (1988) the reference value of the subject's VO2 max. is obtained.
Physical condition (Handgrip Strength) | Through study completion, an average of 1 year
  The test will provide information about the isometric force (kg) that the participant is able to develop with the forearm musculature. For this purpose, a digital dynamometer with manual grip (5030J1, Jamar ®, Sammons Preston, United Kingdom) will be used. Prior to the execution, the instrument will be adjusted according to the age of the player and the length of his/her hand. Two measurements will be taken with each arm, with a one minute rest between them. The participant must hold the dynamometer with the executing hand and the arm extended along the torso, without contacting it, and produce the maximum force possible (Rojas, Vázquez, Sánchez, Banik, & Argáez, 2012; Valdes & Yanci, 2016). Manual grip strength determined by dynamometer is significantly associated with proper cardiovascular health in adolescents, so its analysis is of interest as part of an assessment of global physical fitness (García-Hermoso et al., 2019).
Physical condition (Lower extremity muscle strength) | Through study completion, an average of 1 year
  The countermovement jump test (CMJ) will be used to measure this variable. This test provides information on the explosive strength of the lower body. The CMJ is a vertical jump that begins with the subject in a standing position, followed by knee flexion to a position of approximately 90 degrees, and a rapid extension of the knees to perform a jump in which the maximum height is reached. It should be noted that there is no stop in the knee flexion position since the intention is to take advantage of the explosive elastic reflex energy of the movement. The subjects will perform two repetitions of the jump 2 minutes apart. A MuscleLab force platform (Ergotest Innovation S.A., Norway) will be used to record the data, which will measure the time of flight from the time the subject takes off from the platform to the time the subject re-enters contact with the platform.
Physical condition (Hamstrings Flexibility) | Through study completion, an average of 1 year
  The sit-and-reach test will be used. A 30-centimeter measuring box (Finder Flex-Tester, Novel Products, USA) with a millimeter ruler is required. In the initial position, the subject should be in a seated position, with knees fully extended, feet hip-width apart and soles of the feet perpendicular to the floor and in contact with the box. The subject will be asked to place one hand on top of the other, with the palms of the hands facing downward and the fingers stretched out. The subject will perform a neck flexion to bring the chin to the chest and a trunk flexion with the knees fully stretched and without ballistic movements, trying to reach the greatest possible distance and maintaining the posture for 3 seconds. The distance will be measured in centimeters and the value 0 will correspond to the tangent of the soles of the feet, the values being positive when this distance is exceeded, and negative when it is not reached.
Anthropometric Variables (Height) | Through study completion, an average of 1 year
  To measure height, a SECA measuring rod should be used. Adolescents should stand barefoot with their backs against the measuring rod, heels of their feet together and their gaze straight ahead. Measurements will be obtained in centimeters and will be repeated 2 times for each subject. A third measurement will only be taken if the difference between the first and second measurement is greater than 1%.
Anthropometric Variables (Weight) | Through study completion, an average of 1 year
  A Tanita BC 418-MA Segmental scale (Tanita, Tokyo) will be used to measure body weight. The subject will step on the scale with both feet inside the scale and looking straight ahead, without leaning the body. Values will be obtained in kilograms and two measurements will be carried out on each subject. If the difference between both measurements is greater than 1%, a third measurement will be taken.
Anthropometric Variables (Fat mass) | Through study completion, an average of 1 year
  To obtain the fat mass, it will be necessary to previously measure the triceps, thigh and leg folds, and the waist, hip, relaxed arm, thigh and leg perimeters. For these previous measurements, two measurements will be taken in each subject, and a third measurement will be necessary if the difference between the first two is greater than 5%. Once the values of the previous measurements have been obtained, the fat mass can be calculated using the formula of Slaughter et al. (1988)
Anthropometric Variables (Fat-free mass) | Through study completion, an average of 1 year
  To obtain the fat-free mass, it will be necessary to previously measure the triceps, thigh and leg folds, and the perimeters of the waist, hip, relaxed arm, thigh and leg. For these previous measurements, two measurements will be taken in each subject, and a third measurement will be necessary if the difference between the first two is greater than 5%. Once the values of the previous measurements have been obtained, the-fat free mass can be calculated using the formula of Poortmans et al. (2005)
Anthropometric Variables (BMI) | Through study completion, an average of 1 year
  Previously obtained height and weight measurements will be used to establish the BMI. The formula used will be weight/height^2, and the result will be obtained in kg/m^2. This index is commonly used and is related to metabolic and cardiovascular diseases in adolescents and adults.

CONTACTS AND LOCATIONS:
Overall Officials: Adrián Mateo-Orcajada, MSc, Principal Investigator — Universidad Católica San Antonio
Locations (1):
- Universidad Católica San Antonio, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomez-Cuesta N, Mateo-Orcajada A, Merono L, Abenza-Cano L, Vaquero-Cristobal R. A mobile app-based intervention improves anthropometry, body composition and fitness, regardless of previous active-inactive status: a randomized controlled trial. Front Public Health. 2024 Aug 12;12:1380621. doi: 10.3389/fpubh.2024.1380621. eCollection 2024. PMID 39193194